CLINICAL TRIAL: NCT01335256
Title: An Open-label, Phase I, Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of BAY1000394 Given in a 4 Week on / 2 Week Off Schedule in Subjects With Advanced Malignancies
Brief Title: Clinical Study to Evaluate Safety and Maximum Tolerated Dose of BAY1000394 Given in a 4 Week on / 2 Week Off Schedule in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14856; 2010-019191-79 (EudraCT Number)
Record Dates: First submitted 2011-01-10; First posted 2011-04-14 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Neoplasms
Keywords: Phase I, dose escalation, kinase inhibitor, cyclin-dependent kinase inhibitor, target therapy, small molecule
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY1000394

INTERVENTIONS:
Drug: BAY1000394 — BAY1000394 will be administered orally twice a day (bid) in a 4 week on / 2 week off schedule.

SUMMARY:
Clinical study to determine safety, tolerability, and maximum tolerated dose of BAY1000394 given in 4 week on / 2 week off schedule to patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Subjects with advanced, histologically or cytologically confirmed solid tumors, refractory to any standard therapy, have no standard therapy available, or subjects must have actively refused any treatment which would be regarded standard, and / or if in the judgment of the investigator, experimental treatment is clinically and ethically acceptable
* At least 1 tumor lesion measurable by computer tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST 1.1
* Estimated creatinine clearance 60 mL/min according to Modification of Diet in Renal Disease Study Group (MDRD) formula(2)
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the first dose of study drug
* Subjects with a history of hypertension should be on a stable anti-hypertensive treatment for more than 7 days prior to the first dose of study drug
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study-specific procedures.

Exclusion Criteria:

* Any patient with potentially curable disease will be explicity excluded from enrollment into the study
* Known hypersensitivity to the study drug (active investigational medicinal product or excipients of the preparations) or any agent given in association with this study
* History of cardiac disease: congestive heart failure > NYHA Class II, unstable angina (anginal symptoms at rest), new-onset angina (within the past 3 months prior to study entry), myocardial infarction within the past 3 months prior to study entry, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C(3)
* History of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Symptomatic metastatic brain or meningeal tumors unless the subject is >3 months from definitive therapy, has no evidence of tumor growth on an imaging study within 4 weeks prior to study entry, and is clinically stable with respect to the tumor at the time of study entry. Subjects must not be on acute steroid therapy or taper off steroid therapy (chronic steroid therapy is acceptable provided that the dose is stable for 4 weeks prior to study entry and following screening CT / MRI scan). Subjects with neurological symptoms should undergo a CT / MRI scan of the brain to exclude new or progressive brain metastases. Spinal cord metastasis is acceptable
* Previous or coexisting cancer that is distinct in primary site or histology from the cancer evaluated in this study EXCEPT cervical cancer in-situ, treated basal cell carcinoma, superficial bladder tumors [Ta and Tis], or any cancer curatively treated >3 years prior to study entry
* Anticancer chemotherapy or immunotherapy within 4 weeks of study entry. Mitomycin C or nitrosoureas should not be given within 6 weeks of study entry. Anticancer therapy is defined as any agent or combination of agents with clinically proven anti tumor activity administered by any route with the purpose of affecting the malignancy, either directly or indirectly, including palliative and therapeutic endpoints. Accepted exceptions are bisphosphonates, Luteinizing hormone-releasing hormone (LHRH) agonists for prostate cancer, and mitotane for adrenal carcinoma.
* Radiotherapy to target lesions within 3 weeks prior to the first dose of study drug. Palliative radiotherapy will be allowed as described in Section 6.9 of this protocol. Radiotherapy to the target lesions during study will be regarded as progressive disease
* Use of biological response modifiers, such as granulocyte-colony stimulating factor (G-CSF), within 3 weeks prior to the first dose of study drug. Granulocyte-colony stimulating factor (G-CSF) and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator, however, they may not be substituted for a required dose reduction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events as a measure safety | Up to 3 years or longer if indicated
Maximum tolerated dose: Measured by adverse event profile | Up to 3 years or longer if indicated

SECONDARY OUTCOMES:
Biomarkers evaluation measured by Enzyme-linked immunosorbent assay (ELISA) | Up to 3 years or longer if indicated
Tumor Response evaluation measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to 3 years or longer if indicated
Peak Plasma Concentration (Cmax) of BAY1000394 | Approximately 18 months
Pharmacokinetics parameters will be measured using Peak Plasma Time (tmax) of BAY1000394 | Approximately 18 months
Area under the plasma concentration versus time curve from 0 to tn (AUC(0 tn)) of BAY1000394 | Approximately 18 months
Area under the plasma concentration versus time curve (AUC) of BAY1000394 | Approximately 18 months
Half-life of BAY1000394 | Approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- United States (3):
  - Scottsdale, Arizona
  - St Louis, Missouri
  - Chapel Hill, North Carolina